CLINICAL TRIAL: NCT05233878
Title: Prognostic's Factors of Head and Neck Paragangliomas Evolution
Acronym: PRONO-PARAG
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0295
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-06-30 (Actual); Status verified 2025-06

CONDITIONS: Paraganglioma
Keywords: Cervical paragangliomas
MeSH Terms: conditions — Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort group: Patients over 18 with a confirmed diagnosis of one or multiple cervical paragangliomas
  Interventions: Other: Characterization of a population with cervical paragangliomas

INTERVENTIONS:
Other: Characterization of a population with cervical paragangliomas — Characterization of a population with sporadic or genetically predisposed cervical paragangliomas in order to evaluate : the initial presentation of the PGL, patients management and patients outcome

SUMMARY:
Cervical paragangliomas (HNPG) are rare tumors (0.6% of head and neck tumors) arising from chromaffin tissue, of cervical paraganglia (PGL). The most common locations are carotid body (60% of cases), jugulo-tympanic region and vagal body.

More than 30% are proved to occur in a context of genetic predisposition, more often in young people, and genetic screening is recommended in all patients. Multifocal tumors represent 12% of all HNPG and until 50% of familial forms. Most of HNPG are non-secreting, benign and slow growing tumors, but up to 30% present complications of local growth, and up to 10% can develop distant metastasis that define malignancy since there is no pathological marker.

Historically, surgical treatment was the standard of care but represents nowadays around 50% of the treatment, mostly due to the identification of high morbidity rates. The rate of recurrence is probably around 10% at 5 years. Radiotherapy and active follow-up represent the main therapeutic alternatives.

The standard of care is classically surgical but may expose to important sequelae leading to a review of its primary indication. Indeed, cranial nerve palsies (VII, IX, X, XI and XII) may complicate up to 20% of carotid PGL surgeries and up to 95% of vagal PGL surgeries. They are leading to significant functional sequelae, sometimes requiring recourse to a gastrostomy (4/79 patients operated on in a retrospective cohort). First bite syndrome, Claude Bernard Horner syndrome, baroreceptor failure, xerostomia, and ischemic events complicate 5.8%, 4.9%, 1.9%, 1%, and 1% of surgeries respectively. In a local retrospective study conducted by the Hospices Civils de Lyon on 34 operated cervical PGL, the overall complication rate reached 62%. These complications depend mainly on the location tumor and its size.

Control rate of irradiated HNPG at 5 years from retrospective series seems to be around 90%. They seems also to have a possible better progression-free survival at 15 years than surgery. The tolerance is correct, the risk of induced malignancy is estimed at 1/1000 to 1/2000. Without treatment, 44% of cervical PGL show a significant progression (median follow-up 51 months). Progression is estimated at 0.41 mm/year for jugulo-tympanic PGL and 1.6 mm/year for vagal and carotid PGL.

Currently, there is no clear and robust consensus regarding the follow-up of cervical PGL and the indications for different therapeutic strategies. Data available are represented by retrospective studies only, mostly small in size, with heterogeneous and often inadequate follow-up compared to slow tumor growth.

Thus, this prospective cohort study with a standardized long-term follow-up will allow to characterize the management modalities and the evolution of this population.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 or over
* Patient with a confirmed diagnosis of one or multiple cervical paragangliomas regardless of genetic predisposition without specific therapy
* Patient informed of the study details and who didn't opposed to participate in this research

Exclusion Criteria:

* Patient already treated without initial clinical and radiologic assessment standardized
* Patient already treated with surgery, radiotherapy or systemic therapy for another paraganglioma
* Patient with evolutive disease and life expectancy less than 2 years
* Patient placed under legal protection
* Patient participating in another interventional clinical study that may interfere with the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of one or multiple cervical paragangliomas
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of a population with sporadic or genetically predisposed cervical paragangliomas | 24 months
  Evaluation of the initial presentation of the PGL, patients management and patients outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération d'endocrinologie Hôpital Cardiologique/Groupement Hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No